CLINICAL TRIAL: NCT06197698
Title: A Proof-of-concept Study Evaluating the Microbiota-gut-brain Axis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202112226MINC
Record Dates: First submitted 2023-11-30; First posted 2024-01-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-FDG PET is used as an imaging marker of gut microbiota composition evaluation in PD patients (Other): We will investigate the correlation between 18F-FDC PET bowel uptake and dopamine transporter changes in patients with PD.
  Interventions: Diagnostic Test: F18-FDG, Tc-99m TRODAT-1

INTERVENTIONS:
Diagnostic Test: F18-FDG, Tc-99m TRODAT-1 — In this project, 18F-FDG PET is used as an imaging marker of gut microbiota composition evaluation in PD patients, and the nigrostriatal dopamine system is assessed by Tc-99m TRODAT-1 SPECT.

SUMMARY:
The concept of "Microbiota-gut-brain axis" has long been elucidated. However, only few microbiota-related radionuclide imaging studies have been published. The etiology of physiologic bowel FDG uptake is not fully understood. Some previous studies suggested that bacteria play a role in accumulating FDG and the variability of intestinal FDG activity may rely on a specific type of bacteria in the lumen. It is unclear if FDG transfer from the blood to the bowel lumen through a transcellular or paracellular pathways. The GLUT transporters are known to export glucose from mucosal cells to the blood, but it is doubtful they can also transport in the opposite direction. Therefore, some research speculated the focal or intense FDG uptake might be caused by an increase in intestinal permeability and reflects intestinal barrier impairment.

Gut microbiota compositional changes may affect pathogenesis in patients with Parkinson's disease (PD). A previous hypothesis of PD pointed disease originates in the enteric nervous system and spreads via autonomic neurons to the brain, eventually causing PD. Besides, several studies support the clinical use of Tc-99m TRODAT-1 SPECT in assessing the neurodegenerative status of PD. To date, the correlation between physiologic bowel FDG uptake and dopamine transporter degeneration, as evaluated by either semiquantitative or visual analyses, has never been elucidated.

The objective of this study is to investigate the relationship between the pattern of intestinal FDG activity and Tc-99m TRODAT-1 SPECT images based on the theory of "Microbiota-gut-brain axis".

DETAILED DESCRIPTION:
The key role of gut microbiota in keeping local and systemic homeostasis is termed the "Microbiota-gut-brain axis", which is a complex bidirectional communication system between the gastrointestinal tract and the brain. The hypothalamic-pituitary adrenal (HPA) axis takes part to this bidirectional communication by releasing corticotrophin-releasing factor (CRF), which facilitates the release of adenocorticotrophin hormone (ACTH) from the pituitary, which enters systemic circulation to lead to the release of cortisol from the adrenal glands. Many reports indicating that this hormonal cascade has a significant role in the adjustment of several functions like gastrointestinal transit, visceral sensation and permeability of the intestinal wall.

The etiology of intestinal FDG uptake without pathologic lesions is not fully understood. Tohihara et al. reported physiologic bowel FDG activity at the delayed phase was more than that at the early phase in dual-time images, and postulated FDG secretion was the major cause of physiologic uptake. Franquet et al. reported that physiologic bowel FDG uptake was inhibited by antibiotics, such as rifaximin. Some studies proposed that a specific type of bacteria in the lumen plays a role in gathering FDG, and it explain individual differences in physiologic bowel FDG activity. Previous studies debated about if FDG transfer from the blood to the bowel lumen through a transcellular or paracellular pathways. The GLUT transporters are known to export glucose from mucosal cells to the blood, but it is doubtful they can also transport in the opposite direction. If bowel FDG uptake is associated to intestinal permeability, FDG is likely to migrate through a paracellular pathway because intestinal permeability is adjusted by paracellular tight junction.

There is strong evidence that microbial strains may generate neuroactive molecules such as neurotransmitters, which may interfere with gut and brain functions. Furthermore, gut microbiota compositional changes may affect pathogenesis in patients with Parkinson's disease (PD). A previous hypothesis of PD pointed disease originates in the enteric nervous system and spreads via autonomic neurons to the brain, eventually causing PD. Besides, several studies support the clinical use of Tc-99m TRODAT-1 SPECT in assessing the neurodegenerative status of PD.

To date, no radionuclide imaging studies for correlation between physiologic bowel FDG uptake and dopamine transporter degeneration have been elucidated. The investigators hope to have insight into pathophysiology of PD by investigating the association between the pattern of intestinal FDG activity and Tc-99m TRODAT-1 SPECT images. In addition, research in this field opens the possibility to use neuroactive molecule-producing probiotics as new potential therapeutic tools for patients with PD.

ELIGIBILITY:
Inclusion Criteria:

1. 80 Parkinson's disease patients over 20 years old (the Unified Parkinson's Disease Rating Scale and Hoehn-Yahr Grading Scale are required to provide clinical staging).
2. 20 non-Parkinson's disease patients over 20 years old (control group).
3. Those who are not currently using Metformin, can tolerate fasting for 8 hours, have not used antibiotics within 3 months, and have no obvious intestinal diseases.
4. Subjects and their families agree to join the trial and agree to undergo fluorine-18 deoxyglucose positron imaging (100 subjects will be paid for by research funds) and phosphonium-99m dopamine transporter scan (20 non-Parkinson's patients will be paid for by research funds) syndrome patients) examination.

Exclusion Criteria:

1. Unable to accept positron or single photon angiography such as checking for panic disorder and hemodynamic instability.
2. The possible cancer risk caused by the radiation dose obtained from the experiment cannot be accepted.
3. Pregnant women or women currently breastfeeding.
4. There is a lack of recent unified Parkinson's disease rating scale and Hoehn-Yahr grading scale, making it impossible to know the clinical stage.
5. Those who are currently using Metformin, cannot tolerate fasting for 8 hours, have used antibiotics within 3 months, and have obvious intestinal diseases.
6. The subjects and their families do not agree to join the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Physiological parameter (visual score 1-3) | through study completion, an average of 2 years
  Intestinal FDG uptake classified by visual analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsien Chou, MD, Study Director — NTUH Yunlin branch
Locations (1):
- National Taiwan University Hospital Yunlin branch, Douliu, Taiwan